CLINICAL TRIAL: NCT02002039
Title: Erythropoietin in Perinatal Asphyxia: A Randomized Placebo Controlled Trial
Brief Title: Neuroprotective Role of Erythropoietin in Perinatal Asphyxia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sheri Kashmir Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr.Mushtaq, Professor, Sheri Kashmir Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Erythropoietin 01
Record Dates: First submitted 2013-11-27; First posted 2013-12-05 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Perinatal Asphyxia
Keywords: Perinatal asphyxia; erythropoietin
MeSH Terms: interventions — Erythropoietin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- erythropoietin, perinatal asphyxia, (Active Comparator): Treatment group
  Interventions: Drug: Erythropoietin
- Normal saline, perinatal asphyxia (Placebo Comparator): Normal saline on alternate days for 5 doses starting from first 6 hours of life
  Interventions: Drug: Erythropoietin

INTERVENTIONS:
Drug: Erythropoietin — 500 units /kg /day every other day for 5 doses
  Other Names: erhthropoietin beta

SUMMARY:
Whether Erythropoietin improves the neurological outcomes of neonates with perinatal asphyxia.

DETAILED DESCRIPTION:
will be a randomized trial

ELIGIBILITY:
Inclusion Criteria:

* Babies with severe perinatal asphyxia with moderate to severe HIE in the immediate neonatal period

Exclusion Criteria:

* Babies with congenital malformations
* Small for gestational age babies
* Babies with chromosomal anomalies

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2012-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Death or moderate or severe disability at 18-22 months of age | 18-22 months

SECONDARY OUTCOMES:
Disability | 18-22 months
  Severe disability was defined as GMFCS grade of level 3-5, hearing impairment requiring hearing aids, bilateral cortical visual impairment with no useful vision or Bayley Mental Development Index Score less than 70. Moderate disability was defined as Bayley Mental Developmental Index Score between 70-84 and any one of the following criteria: GMFCS grade of level 2, hearing impairment with no amplification or persistent seizure disorder.
Bayley psychomotor development index | 18-22 months months
Hearing loss at 18-22 months | 18-22 months

CONTACTS AND LOCATIONS:
Overall Officials: Feroz Shaheen, MD, Study Chair — SKIMS; Prof. WAjid Ali, Study Director — SKIMS
Locations (1):
- Sheri-Kashmir Institute of Medical Sciences, Srinagar, Jammu and Kashmir, India

IPD SHARING:
Plan to Share IPD: No